CLINICAL TRIAL: NCT04600648
Title: Sweet Taste Responsiveness in Relation to Insulin, Leptin and Adiposity Among Obese Treatment Seeking Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Carroll M. Harmon, MD PhD, MD, Surgeon-in-Chief and Program Director, University at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00002306
Record Dates: First submitted 2019-08-26; First posted 2020-10-23 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2020-10

CONDITIONS: Pediatric Obesity
Keywords: Leptin; Insulin; Sweet Responsiveness; Weight Loss
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Weight Loss

STUDY DESIGN:
Intervention Model Description: Compare the level of insulin, leptin, and sweet taste sensitivity and perception before and after short term weight loss and bariatric surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight loss with bariatric surgery (Active Comparator): Patients scheduled to undergo bariatric surgery will be tested pre and post bariatric surgery. Interventions to be measured are serum Insulin and leptin levels, sweet taste responsiveness, body fat percentage, and z-BMI
  Interventions: Diagnostic Test: Serum insulin level
- Weight Loss (Active Comparator): Patients to receive lifestyle weight loss treatment will be tested pre and post bariatric surgery. Interventions to be measured are serum Insulin and leptin levels, sweet taste responsiveness, body fat percentage, and z-BMI
  Interventions: Diagnostic Test: Serum Leptin test

INTERVENTIONS:
Diagnostic Test: Serum insulin level — Measure levels before and after weight loss related to bariatric surgery
  Arms: Weight loss with bariatric surgery
Diagnostic Test: Serum Leptin test — Measure levels before and after weight loss related to lifestyle change weight loss
  Arms: Weight Loss

SUMMARY:
This study will explore whether a relationship exists between insulin and leptin resistance, sweet taste responsiveness, and adiposity.

DETAILED DESCRIPTION:
Compared to healthy weight peers, some reports have shown that they are less sensitive to, or perceptive of, sucrose solutions and sweet foods, whereas others have observed the opposite pattern of findings or no difference at all. Among those seeking weight loss treatment, one investigation found perception and preferences for sweet taste remained unchanged after weight loss, and another observed a decreased ability to distinguish sweet taste from other taste solutions. Given these discrepancies in the literature, the proposed study will explore whether a relationship exists between insulin and leptin resistance, sweet taste responsiveness, and adiposity.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Children's Healthy Weigh of Buffalo
* ages of 8-14

If enrolled in the bariatric arm:

• must be scheduled for bariatric surgery prior to enrollment

Exclusion Criteria:

* Patients unable to get labs drawn at a Kaleida facility
* Severe hay fever or seasonal allergies within 2 weeks of enrollment
* smoker or are exposed to second-hand smoke at home,
* has been dieting to lose weight within the past 6 months of enrollment
* currently taking any prescription medications that can influence taste or small functions or are pregnant.
* pregnancy
* Bariatric arm patients will be excluded if they fail to have the surgery.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Higher insulin and leptin levels will be associated with lower sweet taste sensitivity and perception, and higher body fat percentage and z-BMI | to be measured at 6 months
  insulin and leptin levels will be measured at various time points in an attempt to identify if there is a change is taste senses associated with specific variables be associated with lower sweet taste